CLINICAL TRIAL: NCT04173819
Title: Safety and Pharmacokinetics of the Combination Broadly Neutralizing Antibodies, 3BNC117-LS-J and 10-1074-LS-J, in Healthy American and African Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Fred Hutchinson Cancer Center (Other); Rockefeller University (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IAVI C100
Record Dates: First submitted 2019-11-13; First posted 2019-11-22 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blind, placebo-controlled Phase 1/2 study intended to evaluate the safety and pharmacokinetics of 10-1074-LS-J and 3BNC117-LS-J, alone or in combination, in healthy HIV-uninfected individuals.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Group 1 (Experimental): Single Agent, abdominal subcutaneous injection, 10:2 ratio for Ab:placebo
  Interventions: Biological: 3BNC117-LS-J; Biological: Placebo
- Group 2 (Experimental): Single agent, abdominal subcutaneous injection 10:2 ratio for Ab:placebo
  Interventions: Biological: 10-1074-LS-J; Biological: Placebo
- Group 3 (Experimental): Single agent intravenous injection 10:2 ratio for Ab:placebo
  Interventions: Biological: 3BNC117-LS-J; Biological: Placebo
- Group 4 (Experimental): Single agent intravenous injection 10:2 ratio for Ab:placebo
  Interventions: Biological: 10-1074-LS-J; Biological: Placebo
- Group 5 (Experimental): Combined agent intravenous injection 10:2 ratio for Ab:placebo
  Interventions: Biological: Combination 3BNC117-LS-J and 10-1074-LS-J; Biological: Placebo
- Group 6 (Experimental): Subcutaneous injection combined ratio 1 with loading dose 30:3 ratio of Ab:Placebo
  Interventions: Biological: Combination 3BNC117-LS-J and 10-1074-LS-J Ratio 1; Biological: Placebo
- Group 7 (Experimental): Subcutaneous injection in abdomen combined ratio 2 with loading dose 30:3 ratio of Ab:Placebo
  Interventions: Biological: Combination 3BNC117-LS-J and 10-1074-LS-J Ratio 2; Biological: Placebo
- Group 8 (Experimental): Subcutaneous injection in abdomen combined ratio 3 with loading dose 30:3 ratio of Ab:Placebo
  Interventions: Biological: Combination 3BNC117-LS-J and 10-1074-LS-J Ratio 3; Biological: Placebo
- Group 9 (Experimental): Subcutaneous injection in abdomen combined ratio 2 without loading dose 30:3 ratio of Ab:Placebo
  Interventions: Biological: Combination 3BNC117-LS-J and 10-1074-LS-J Ratio 2; Biological: Placebo
- Group 10 (Experimental): Subcutaneous injection in arm combined ratio 2 without loading dose 30:3 ratio of Ab:Placebo
  Interventions: Biological: Combination 3BNC117-LS-J and 10-1074-LS-J Ratio 2; Biological: Placebo

INTERVENTIONS:
Biological: 3BNC117-LS-J — 300mg
  Arms: Group 1; Group 3
Biological: 10-1074-LS-J — 300mg
  Arms: Group 2; Group 4
Biological: Combination 3BNC117-LS-J and 10-1074-LS-J — 30mg/kg of each
  Arms: Group 5
Biological: Combination 3BNC117-LS-J and 10-1074-LS-J Ratio 1 — Total ~300 mg (< 2.5 ml) combined of 3BNC117-LS-J and 101074-LS-J - Dosage ratios chosen will be those considered worthy of further investigation based on the safety and preliminary PK observed in groups 1-2
  Arms: Group 6
Biological: Combination 3BNC117-LS-J and 10-1074-LS-J Ratio 2 — Total ~300 mg (< 2.5 ml) combined of 3BNC117-LS-J and 101074-LS-J - Dosage ratios chosen will be those considered worthy of further investigation based on the safety and preliminary PK observed in groups 1-2
  Arms: Group 10; Group 7; Group 9
Biological: Combination 3BNC117-LS-J and 10-1074-LS-J Ratio 3 — Total ~300 mg (< 2.5 ml) combined of 3BNC117-LS-J and 101074-LS-J - Dosage ratios chosen will be those considered worthy of further investigation based on the safety and preliminary PK observed in groups 1-2
  Arms: Group 8
Biological: Placebo — 0.9% Saline
  Arms: Group 3; Group 4; Group 5
Biological: Placebo — Buffer Solution
  Arms: Group 1; Group 10; Group 2; Group 6; Group 7; Group 8; Group 9

SUMMARY:
This is a Phase 1/2 study to evaluate the safety, tolerability, and pharmacokinetics of two broadly neutralizing monoclonal human antibodies (bNAbs), 3BNC117-LS-J, which targets the CD4 binding site on HIV-1 envelope protein, and 10-1074-LS-J which targets the V3 loop of HIV-1 envelope protein. The hypothesis is that the two antibodies will be safe for healthy HIV-1 uninfected adults when co-administered subcutaneously or intravenously and, after subcutaneous administration in the optimal ratio, each antibody will maintain serum levels >10 µg/ml for at least 3 months in HIV-uninfected participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female individuals, as assessed by a medical history, physical exam, and laboratory tests
* At least 18 years of age on the day of screening and have not reached their 46th birthday on the day of the first administration
* Willing to undergo HIV testing, risk reduction counseling and receive HIV test results; committed to maintaining low-risk behavior for the trial duration
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study
* All male and female participants of reproductive potential who are engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception from enrollment until 9 months after the last administration
* Willing to forgo donations of blood, or any other tissues during the study following confirmation of study eligibility and, for those who test HIV-positive due to antibody-induced seropositivity, until the anti-HIV antibody titers become undetectable on HIV tests used in the community

Exclusion Criteria:

* Confirmed HIV infection
* Reported risk for HIV infection within 6 months prior to investigational product administration, as defined by: Unprotected sexual intercourse with a known HIV-infected person, a partner known to be at high risk for HIV infection and/or a casual partner (i.e. no continuing established relationship), engaged in sex work, frequent excessive daily alcohol use or frequent binge drinking or any other use of illicit drugs, history of newly-acquired syphilis, gonorrhea, non-gonococcal urethritis, HSV-2, chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B or hepatitis C, three or more sexual partners
* Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the investigator makes the participant unsuitable for participation in the study
* Infectious disease diagnosis: Hepatitis B infection as measured by HbsAg and/or PCR, Hepatitis C infection (US: HCV RNA positive, or interferon-alpha treatment for hepatitis C infection in the past year, or interferon-alpha-free treatment for hepatitis C infection completed in the past 6 months; Africa: HCV Ab positive and/or PCR positive), active syphilis (positive RPR confirmed by TPHA)
* Receipt of blood transfusion or blood-derived products within the previous 3 months
* Participation in another clinical trial of an investigational product currently, within the previous 3 months or expected participation during this study (Concurrent participation in an observational trial not requiring blood or tissue sample collection is not an exclusion)
* Psychiatric condition that compromises safety of the participant and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
* Body mass index (BMI) >40
* Active tuberculosis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
1. Proportion of participants with solicited and treatment-related unsolicited adverse events and their duration. | 92 Weeks
Proportion of participants with serious adverse events (SAEs) throughout the study period that are considered related to investigational product and their duration. | 92 Weeks
Serum concentration of each antibody in each group at multiple timepoints along with participant characteristics (e.g. sex, weight, and BMI) | 92 Weeks
The ratio of 3BNC117-LS-J to 10-1074-LS-J that, when injected SC, will maintain similar levels of each bNAb at steady state. | 92 Weeks

SECONDARY OUTCOMES:
Serum concentration of anti-3BNC117-LS-J antibodies in each group at multiple timepoints. | 92 Weeks
Serum concentration of anti-10-1074-LS-J antibodies in each group at multiple timepoints. | 92 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Study Chair — Rockefeller University
Locations (9):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - The Rockefeller University, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Kenya (2):
  - Partners in Health Research and Development, Thika, Kiambu County
  - Kenya AIDS Vaccine Initiative - Institute of Clinical Research, Nairobi
- Center for Family Health Research, Kigali, Rwanda
- Wits Reproductive Health and HIV Institute, Johannesburg, South Africa
- Uganda (2):
  - Uganda Virus Research Institute, Entebbe
  - Infectious Diseases Institute Kasangati, Kampala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://iavi.org